CLINICAL TRIAL: NCT00021632
Title: Pharmacokinetic Evaluation of the Effects of Ribavirin (RBV) on Zidovudine (ZDV) or Stavudine (d4T) Triphosphate (TP) Formation
Brief Title: Effects of Ribavirin on Zidovudine or Stavudine
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5092s; AACTG A5092s; ACTG A5092s; 10919 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2001-07-26; First posted 2001-08-31 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; Hepatitis C
Keywords: Ribavirin; Drug Interactions; Drug Therapy, Combination; Zidovudine; Stavudine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Pharmacokinetics; Area Under Curve
MeSH Terms: conditions — HIV Infections; Hepatitis C

SUMMARY:
The purpose of this study is to see how treatment of hepatitis C (HCV) patients with ribavirin (RBV) affects the anti-HIV drugs stavudine (d4T) or zidovudine (ZDV).

Studies have shown that RBV may interfere with the action of ZDV and d4T. There is little information about the way these drugs interact in the body. This study will examine how the drug RBV affects levels of ZDV or d4T in patients who are currently on stable anti-HIV therapy.

DETAILED DESCRIPTION:
RBV, a nucleoside analogue, is used for the treatment of hepatitis C virus (HCV) in alliance with interferon-alfa 2a/2b in patients with HIV-1. The mechanism of action of RBV has led to in vitro studies examining the agonism/antagonism in efficacy occurring when used in combination with nucleoside reverse transcriptase inhibitors (NRTIs). The primary objective of the pharmacology component of this current study will be the evaluation of the effect of RBV on the intracellular activation of ZDV or d4T owing to the reported antagonism observed in vitro.

Pharmacokinetic (PK) evaluations for plasma ZDV or d4T and intracellular ZDV or d4T and measurements of their triphosphate anabolites are performed before initial RBV dosing (within 2 weeks of visit) and 8 weeks after RBV administration. Thymidine triphosphate (TTP) concentrations also are quantitated to permit estimation of the ratio of active drug to endogenous triphosphate concentrations.

For entry, prior to RBV dosing, blood samples are collected within 2 hours prior to the ZDV or d4T dose and then at Hours 1, 4, and 8 post dosing. Following the entry PK blood draws, patients initiate RBV treatment within 2 weeks of the first PK study day.

For the Week 8 evaluation (measured as 8 weeks following initiation of RBV), blood samples are collected prior to the ZDV or d4T dose and then at Hours 1, 4, and 8 post dosing.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years of age.
* Have written consent from parent or guardian if under 18 years of age.
* Have HIV infection.
* Have been receiving ZDV or d4T for at least 4 weeks prior to study entry.
* Are planning to receive RBV-containing hepatitis treatment through their doctor or through coenrollment in another ACTG protocol within 2 weeks following entry into the study.
* Have not received RBV for at least 6 months prior to study entry if they were previously treated with RBV.
* Weigh more than 110 pounds (50 kg).

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant.
* Use rifampin, rifabutin, pyrazinamide, isoniazid, ganciclovir, or hydroxyurea within 14 days of study entry.
* Abuse alcohol or drugs. Patients in methadone programs may participate.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Aweeka, Study Chair
Locations (6):
- United States (6):
  - UCLA CARE Ctr, Los Angeles, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Willow Clinic / Stanford Univ, Stanford, California
  - Johns Hopkins Hosp, Baltimore, Maryland
  - MetroHealth Medical Center, Cleveland, Ohio

REFERENCES:
- [Result] Aweeka FT, Kang M, Yu JY, Lizak P, Alston B, Chung RT; AIDS Clinical Trials Group 5092s Study Team. Pharmacokinetic evaluation of the effects of ribavirin on zidovudine triphosphate formation: ACTG 5092s Study Team. HIV Med. 2007 Jul;8(5):288-94. doi: 10.1111/j.1468-1293.2007.00472.x. PMID 17561874